CLINICAL TRIAL: NCT06374290
Title: Open-label Pilot Study of Injectable Naltrexone and Oral Bupropion Among Cigarette Smokers With Schizophrenia
Brief Title: Study of Injectable Naltrexone and Oral Bupropion Among Cigarette Smokers With Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit eligible participants and expiration of study medication.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jin Ho Yoon, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-24-0024
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation
Keywords: schizophrenia spectrum disorder
MeSH Terms: conditions — Smoking Cessation | interventions — Naltrexone; vivitrol; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Naltrexone (Vivitrol); Drug: Bupropion

INTERVENTIONS:
Drug: Naltrexone (Vivitrol) — At week 1 the Nurse Practitioner will administer extended-release naltrexone via intramuscular gluteal injection supplied as a standard single-use kit containing 380-mg vial of Vivitrol microspheres. Only one naltrexone injection will be administered over the course of the study
Drug: Bupropion — Oral bupropion will be titrated to 450 mg over the course of 3 days. One week's supply of the study medication will be dispensed at each visit. Cell-phone assisted remote observation of medication adherence (CAROMA) will be used to assess compliance. Following Week 3, participants will be provided with enough pills to titrate the dose of bupropion over a period of 4 days. Therefore, participants will receive bupropion pills 3 weeks plus 4 additional days to titrate down the dose.

SUMMARY:
The purpose of this study is to assess the feasibility and safety of injectable naltrexone (NTX;380 mg) in conjunction with oral bupropion (BUP; 450 mg daily)NTX-BUP administration among individuals with schizophrenia spectrum disorders that smoke cigarettes and to evaluate change on smoking-related measures and symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* fluent in English;
* Diagnosed with schizophrenia spectrum disorder that is currently stable;
* Report regular cigarette smoking, average cigarette per day ≥ 5 in the past 4 weeks, and present a breath CO≥10 ppm.
* Meet subjective and objective (urinary drug screen) measures of non-opioid use.
* If female, present a negative pregnancy test, not be currently breast feeding, and agree to use acceptable birth control methods and receive periodic pregnancy tests during the course of the study.
* Able to give written informed consent
* Obtain an Evaluation to Sign Consent (ESC) score above 10.

Exclusion Criteria.

* Have suicidal or homicidal ideation requiring immediate attention.
* Previous use of bupropion or naltrexone in the past 30 days.
* Currently enrolled in treatment for tobacco use.
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5 )criteria for alcohol and other substance use disorders excluding nicotine and marijuana.
* Report a history of epilepsy, seizure disorder or condition increasing risk of seizure, or head trauma with neurological sequelae.
* Have a current eating disorder.
* Be medically unstable or taking medications that are contraindicated with using naltrexone or bupropion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by the percentage of participants that enroll in the study | end of treatment (week 3)
Percentage of participants that complete 3 weeks of treatment | end of treatment (week 3)
Safety as assessed by the percentage of participants that show no serious adverse events | end of treatment (week 3)

SECONDARY OUTCOMES:
Change in number of cigarettes smoked per day (CPD) | Baseline, end of treatment (week 3)
Change in smoking urges as assessed by the Questionnaire on Smoking Urges (QSU) | Baseline, end of treatment (week 3)
  This is a 10 item questionnaire and each is cored from 0(strongly disagree) to 10(strongly agree) for a maximum score of 100, higher score indicating more smoking urge
Reduction in number of cigarettes consumed when price is at 0 as assessed by the Cigarette Purchasing Task (CPT) | Baseline, end of treatment (week 3)
  This will utilize a hypothetical purchasing task, which will assess hypothetical purchase and consumption of cigarettes as a function of increasing cigarette price.
Change in psychiatric symptoms as assessed by the score on the Brief Psychiatric Rating Scale (BPRS) | Baseline, end of treatment (week 3)
  This is an 18 item questionnaire and each is scores from 1 (not present) to 7 (extremely severe),with a total score between 18 and 126, higher number indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jin H Yoon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No